CLINICAL TRIAL: NCT01596283
Title: A Prospective Randomized Controlled Clinical Trial of Standard Compared to Goal-directed Perioperative Fluid Management (GDT) for Patients Undergoing Liver Resection
Brief Title: Clinical Trial of Standard Versus Goal-Directed Perioperative Fluid Management (GDT) for Patients Undergoing Liver Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-056
Record Dates: First submitted 2012-04-30; First posted 2012-05-10 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2016-05

CONDITIONS: Liver Cancer
Keywords: Perioperative Fluid Management; liver resection; 12-056
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Standard fluid management (Active Comparator): Prospective single-blinded randomized trial. Eligible patients will be consented for the trial prior to surgery. However randomization will not occur until the operating room. After the liver has been resected, intraoperative randomization will be done by envelopes.
  Interventions: Procedure: Standard fluid management
- Goal directed fluid therapy (Active Comparator): Prospective single-blinded randomized trial. Eligible patients will be consented for the trial prior to surgery. However randomization will not occur until the operating room. After the liver has been resected, intraoperative randomization will be done by envelopes.
  Interventions: Device: Goal directed fluid therapy with the Edwards EV1000 system

INTERVENTIONS:
Procedure: Standard fluid management — The patient will receive standard fluid management
  Arms: Standard fluid management
Device: Goal directed fluid therapy with the Edwards EV1000 system — This arm will have fluid therapy guided by the Edwards EV1000 system.
  Arms: Goal directed fluid therapy

SUMMARY:
The purpose of this study is to help us learn what is the best amount of fluid to administer to patients during liver surgery. Patients will receive either an amount for this surgery based on weight, blood pressure, heart rate and urine output or an amount guided by a computerized system (FloTrac) that helps doctors know how much fluid each patient needs. The FloTrac calculates the amount of fluid patients needs on a minute-to-minute basis, based on real time information like blood pressure, pulse and the ability of the heart and blood vessels to maintain normal vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years old or greater) who are able to provide informed consent.
* Patients who undergo an open, elective liver resection. Including those initially approached laparoscopically but converted to an open resection and those undergoing additional procedures.

Exclusion Criteria:

* Active coronary disease.
* Patients with a history of coronary disease will be eligible if they have had a cardiac stress study showing no reversible ischemia and normal LV function within 3 months of operation.
* Active symptomatic cerebrovascular disease.
* Active congestive heart failure and ejection fraction <35%.
* Active severe restrictive or obstructive pulmonary disease and resting SpO2 <90%.
* Active renal dysfunction (Cr >1.8)
* Abnormal coagulation parameters (INR > 1.8 not on Coumadin, or platelet count < 100,000 per mcL)
* Presence of active infection including HIV
* Patients with active atrial fibrillation or flutter.
* Preoperative hypoalbuminemia (Albumin < 2g/dl).
* Female patients who are pregnant (female patients of child-bearing potential must have a negative serum pregnancy test ≤ 14 days prior to surgery or 15 to 30 days prior to surgery with a negative urine pregnancy test the morning of surgery).
* Presence of ascites.
* BMI > 45 or <17

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2012-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Fischer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Correa-Gallego C, Tan KS, Arslan-Carlon V, Gonen M, Denis SC, Langdon-Embry L, Grant F, Kingham TP, DeMatteo RP, Allen PJ, D'Angelica MI, Jarnagin WR, Fischer M. Goal-Directed Fluid Therapy Using Stroke Volume Variation for Resuscitation after Low Central Venous Pressure-Assisted Liver Resection: A Randomized Clinical Trial. J Am Coll Surg. 2015 Aug;221(2):591-601. doi: 10.1016/j.jamcollsurg.2015.03.050. Epub 2015 Apr 7. PMID 26206652
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Goal-directed Therapy (GDT) After Liver Resection: Patients who undergo an open, elective liver resection, Including those initially approached laparoscopically but converted to an open resection and those undergoing additional procedures. Goal-directed therapy (GDT) embodies a number of physiologic strategies to achieve an ideal fluid balance and avoid the consequences of over- or under-resuscitation.
- Standard Perioperative Resuscitation After Liver Resection: Patients who undergo an open, elective liver resection, Including those initially approached laparoscopically but converted to an open resection and those undergoing additional procedures.
Period: Overall Study
Arm/Group | Goal-directed Therapy (GDT) After Liver Resection | Standard Perioperative Resuscitation After Liver Resection
Started | 69 | 66
Completed | 69 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Goal-directed Therapy | Standard Perioperative Resuscitation | Total
Number analyzed (Participants) | 69 | 66 | 135
Age, Continuous [Median (Standard Deviation); unit: years] | 55 (13) | 58 (14) | 57 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 39 | 75
  Male | 33 | 27 | 60
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69 | 66 | 135

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Complications
Description: The incidence of overall 30-day postoperative complications will be recorded. These are defined in the MSKCC Adverse Events Program and organized by categories reflecting organ systems and further subdivided into specific complications within those and graded.
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Fluid Management | Goal Directed Fluid Therapy
Number analyzed (Participants) | 66 | 69
Participants
  30-day survival | 42 | 45
  30-day overall morbidity | 24 | 24

2. Secondary Outcome: Low Cardiac Output Time
Description: Assess the impact of GDT compared to standard fluid therapy on the total time patients experience low cardiac output perioperatively
Time Frame: Up to the first 24 postoperative hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard Fluid Management | Goal Directed Fluid Therapy
Number analyzed (Participants) | 66 | 69
minutes | 21 (113) | 12 (48)

3. Secondary Outcome: Total Volume of Fluid Used Perioperatively
Description: Assess the impact of GDT compared to standard fluid therapy on the total volume of fluid given intraoperatively
Time Frame: Up to the first 72 hours postoperatively
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Goal-directed Therapy (GDT) After Liver Resection | Standard Perioperative Resuscitation After Liver Resection
Number analyzed (Participants) | 69 | 66
liter | 2.0 (1.1) | 2.9 (1.0)

4. Secondary Outcome: Total Volume of Fluid Used Postoperatively
Description: Postoperative fluid volume
Time Frame: Postoperatively for the total admission time, up to 8 days
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Goal-directed Therapy (GDT) After Liver Resection | Standard Perioperative Resuscitation After Liver Resection
Number analyzed (Participants) | 69 | 66
liter | 0.9 (0.6) | 1.0 (0.5)

5. Secondary Outcome: Postoperative Length of Stay
Description: Assess the impact of GDT compared to standard fluid therapy on net fluid balance for the total admission time
Time Frame: Postoperatively for the total admission time, up to 8 days
Measure: Median (Full Range); unit: days
Arm/Group | Goal-directed Therapy (GDT) After Liver Resection | Standard Perioperative Resuscitation After Liver Resection
Number analyzed (Participants) | 69 | 66
days | 7 [6 to 8] | 6 [5 to 8]

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Standard Fluid Management | Goal Directed Fluid Therapy
All-Cause Mortality (participants affected / at risk) | 0/66 | 3/69
Serious Adverse Events (participants affected / at risk) | 23/66 | 46/69
Other Adverse Events (participants affected / at risk) | 66/66 | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Fluid Management (N=66) | Goal Directed Fluid Therapy (N=69)
Intra-abdominal infection or abscess (Infections and infestations) | 9 | 13
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Wound infection (Infections and infestations) | 1 | 1
Liver dysfunction/failure (Hepatobiliary disorders) | 0 | 2
Non-infected intra-abdominal/intra-thoracic fluid collection (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Biliary anastomotic leak (Hepatobiliary disorders) | 1 | 2
Biloma (Hepatobiliary disorders) | 1 | 2
Hemorrhage (Blood and lymphatic system disorders) | 0 | 1
Renal Failure (Renal and urinary disorders) | 1 | 3
Sepsis (Infections and infestations) | 1 | 2
Ascites (Gastrointestinal disorders) | 5 | 8
Mortality (General disorders) | 0 | 2
Thromboembolic Event (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Fluid Management (N=66) | Goal Directed Fluid Therapy (N=69)
Intra-abdominal infection of abscess (Infections and infestations) | 10 | 13
Wound infection (Infections and infestations) | 7 | 5
Liver dysfunction/failure (Hepatobiliary disorders) | 1 | 4
Non-infeccted intra-abdominal/intra-thoracic fluid collection (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Biliary anastomotic leak (Hepatobiliary disorders) | 2 | 3
Biloma (Hepatobiliary disorders) | 1 | 3
Hemorrhage (Blood and lymphatic system disorders) | 0 | 3
Renal Failure (Renal and urinary disorders) | 1 | 3
Mortality (General disorders) | 0 | 2
Alanine aminotransferase increased (Investigations) | 66 | 69
Aspartate aminotransferase increased (Investigations) | 66 | 69
Hyperglycemia (Metabolism and nutrition disorders) | 66 | 69
Hypoalbuminemia (Metabolism and nutrition disorders) | 66 | 69
Apnea or Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 3 | 2
Bile duct injury (Injury, poisoning and procedural complications) | 0 | 1
Bowel perforation, necrosis (Gastrointestinal disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Clostridium difficile colitis (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Fascial dehiscence or evisceration (Musculoskeletal and connective tissue disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Foreign body infection (Infections and infestations) | 0 | 2
Fungal infection (Infections and infestations) | 0 | 1
Hepatic arterial infusion pump dysfunction (Hepatobiliary disorders) | 2 | 1
Ileus, paralytic (Gastrointestinal disorders) | 3 | 2
Pneumonia (Infections and infestations) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolus (Vascular disorders) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Small bowel obstruction (Gastrointestinal disorders) | 1 | 0
Splenic injury (Injury, poisoning and procedural complications) | 1 | 0
Supraventricular arrhythmia (Cardiac disorders) | 1 | 1
Vascular thrombosis (Vascular disorders) | 1 | 2
Wound breakdown (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-05-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT01596283/Prot_SAP_000.pdf